CLINICAL TRIAL: NCT03663959
Title: Intermediate-term Outcomes of Laparoscopic Pectopexy and Vaginal Sacrospinous Fixation: A Comparative Study
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, bahar sarıibrahim astepe, obstetrics and gynecology specialist, Kocaeli Derince Education and Research Hospital
Other Study IDs: KOCAELİe-14101
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Laparoscopic Pectopexy and Vaginal Sacrospinous Fixation
Keywords: Outcomes; Pectopexy; Sacrospinous ligament fixation; Prolapse surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaginal Sacrospinous Fixation group: Women who had vaginal sacrospinous fixation procedure with Dr.Aksakal's Desta suture carrier in our clinic between January 2014 and June 2018.
  Interventions: Procedure: vaginal sacrospinous fixation procedure with dr.Aksakal's desta suture carrier
- Laparoscopic Pectopexy Group: Women who had Laparoscopic Pectopexy procedure in our clinic between January 2014 and June 2018
  Interventions: Procedure: Laparoscopic Pectocolpopexy procedure

INTERVENTIONS:
Procedure: vaginal sacrospinous fixation procedure with dr.Aksakal's desta suture carrier — A right sacrospinous fixation using Dr. Aksakal's Desta suture carrier with two permanent sutures that combined the sacrospinous ligament and vaginal cuff fascia was done. The Desta suture carrier was developed for deep pelvic surgery, and the suture depth can be easily adjusted. After the vaginal hysterectomy, under the vaginal cuff mucosa, we created a tunnel through the spinous process with a straight tool. After passing the rectovaginal pillars, the perirectal space was entered and the ischial spine was palpated. With the help of an index finger placed on the spinous process, we placed two permanent sutures 1.5-2 cm medial to the spinous process on the sacrospinous ligament and iliococcygeus muscle complex using the Desta suture carrier. Next, permanent sutures were combined with the pubocervicovaginal and rectovaginal fascia under the vaginal cuff mucosa.
  Groups: Vaginal Sacrospinous Fixation group
Procedure: Laparoscopic Pectocolpopexy procedure — First, the peritoneal layer above and lateral to the bladder was opened parallel to the round ligament toward the pelvic side wall on the right side. Then, with the guidance of the obliterated umbilical artery, lateral to the obliterated umbilical artery and medial to the external iliac vein, the iliopectineal ligament was found . At this point, a segment of approximately 3-4 cm2 was formed, exposing the iliopectineal (Cooper's) ligament. In this area, behind the obliterated umbilical artery, the obturator nerve could be seen, and special care was given not to make contact with the nerve. The same area on the left side was prepared using the same steps. Then, anterior part of the vaginal cuff was prepared for mesh fixation. Bilaterally, the ends of a polypropylene monofilament mesh (1,5x15 cm) were fixed to the iliopectineal ligament with nonabsorbable polypropylene or polyester sutures . The vaginal cuff was elevated to POP-Q level 0-1.
  Groups: Laparoscopic Pectopexy Group

SUMMARY:
Forty-three women who had vaginal sacrospinous fixations using Dr. Aksakal's Desta suture carrier and 36 women who had laparoscopic pectopexies between January 2014 and June 2018 at H.S.U Kocaeli Derince Training and Research Hospital Gynecology and Obstetrics clinic were re-examined between 15 June and 30 December 2018 gynecologically.

DETAILED DESCRIPTION:
Forty-three women who had vaginal sacrospinous fixations using Dr. Aksakal's Desta suture carrier and 36 women who had laparoscopic pectocolpopexies were re-examined 7 to 43 months after surgery. All of the women had undergone surgery for stage 2 or greater uterovaginal or vaginal vault prolapse according to the Pelvic Organ Prolapse Quantification (POP-Q) system.

All of the patients received telephone calls and were invited for a gynecological re-examination. All but one patient in the vaginal surgery group came in for a gynecological control. We conducted a phone interview with the one patient not agreeing to come to the control, and we learned that she had a relapse 6 months after the operation. She underwent another prolapse surgery at a different hospital. She described her postsurgical complaints, and we noted that she was unsatisfied with the surgery. In the postoperative re-evaluation between 15 June and 30 December 2018, all of the women were examined in the lithotomy position for apical, anterior, and posterior compartment descensus. Stage 2 or greater apical descensus or a cystocele or rectocele according to the POP-Q system were accepted as postoperative relapses. All of the patients answered the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) and Prolapse Quality of Life (P-QOL) questionnaire. All of the women were asked about de novo urge urinary incontinence and de novo stress urinary incontinence. In addition, each patient's satisfaction with the surgery was asked and recorded.

ELIGIBILITY:
Inclusion Criteria:

Those patients with stage 2 or greater uterovaginal/vaginal cuff prolapses according to the POP-Q system underwented to surgery (vaginally or laparoscopically) between January 2014 and June 2018 were included to the study.

Exclusion Criteria:

Women who had surgeries for malignancy suspicion or pelvic inflammatory disease and women with pectouteropexy procedure were not included into the study.

Ages: 45 Years to 81 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women who had undergone uterovaginal or vaginal vault prolapse surgery ( vaginal sacrospinous fixation /laparoscopic pectopexy procedures ) between January 2014 and June 2018 at the H.S.U. Kocaeli Derince Education and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Apical descensus relapse rate | 7-43 months after surgery
  The ratio of women with stage 2 or greater vaginal cuff prolapsus according to the Pelvic Organ Prolapse Quantification (POP-Q) system to all women

SECONDARY OUTCOMES:
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) | 7-43 months after surgery
  The PISQ-12 is a self-adminestered questionnaire that evaluates sexual function of women with pelvic organ prolapse or urinary incontinence. The questionnaire has 12 items. Other than the first 4 questions that are scored from 4 to 0, all questions are scored from 0 to 4. The total score is calculated with totaling the score of each question. The maximum score is 48. Higher scores show good sexual functioning of women.
Prolapse Quality of Life (P-QOL) | 7-43 months after surgery
  The P-QOL questionnaire evaluates the impact of urogenital prolapsus on quality of life in women. The questionnaire has nine items, each of has 4-point scoring system and a total score of 0-100. A high total score indicates worsening of quality of life of women with pelvic organ prolapsus.
De novo central or lateral defect cystocele rate | 7-43 months after surgery
  The ratio of women with stage 2 or greater central or lateral defect cystocele according to the Pelvic Organ Prolapse Quantification (POP-Q) system to all women
De novo rectocele rate | 7-43 months after surgery
  The ratio of women with stage 2 or greater rectocele according to the Pelvic Organ Prolapse Quantification (POP-Q) system to all women
Satisfied with surgery rate | 7-43 months after surgery
  The ratio of women satisfied with surgery to all women
De novo stress urinary incontinence rate | 7-43 months after surgery
  The ratio of women with de novo stress urinary incontinence to all women
De novo urge urinary incontinence rate | 7-43 months after surgery
  The ratio of women with de novo urge urinary incontinence to all women

CONTACTS AND LOCATIONS:
Overall Officials: bahar sarıibrahim astepe, Principal Investigator — H.S.U Kocaeli Derince Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Bahar Sarıibrahim Astepe, Kocaeli
  - S.B.U Kocaeli Derince Education and Research Hospital, Kocaeli

IPD SHARING:
Plan to Share IPD: No
The investigators do not prefer to share the study plan and records.